CLINICAL TRIAL: NCT03325829
Title: Diverticular Disease Register (REMAD)
Brief Title: Registro Malattia Diverticolare (Registry of Diverticular Disease)
Acronym: REMAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattia Diverticolare (Other)
Responsible Party: Principal Investigator, ROSARIO CUOMO, Associate Professor of Gastroenterology, Gruppo Italiano Malattia Diverticolare
Other Study IDs: REMAD Registry
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Diverticulum, Colon; Diverticulitis
Keywords: Registry; Diverticular Disease; Diverticulitis; Uncomplicated Diverticular Disease
MeSH Terms: conditions — Diverticulum, Colon; Diverticulitis; Diverticular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with colonic diverticula: No interventional study

SUMMARY:
To determine the clinical characteristics and risk factors for the onset of diverticular disease and its complications in the Italian population.

DETAILED DESCRIPTION:
Diverticulosis and diverticular disease present a high prevalence rate in the world population, especially in the Western world. Diverticulosis of the colon is an extremely common condition in industrialized countries and its prevalence rate increases with age, and exceeds 60% in patients aged over eighty. Although the course of diverticulosis is normally free of symptoms and complications, about 15% of patients develop symptoms often undistinguishable from those of the irritable bowel syndrome, such as abdominal pain, bowel disorders and bloating. About 5% of patients with diverticular disease develop an episode of uncomplicated acute diverticulitis with abdominal symptoms accompanied in some cases by systemic symptoms, such as fever or malaise and laboratory evidence of activation of the inflammatory process. In a minority of these cases, the patient suffers major complications such as the development of abscesses, fistulae, haemorrhage or stenosis (1).

The pathogenesis of diverticulosis and diverticular disease remains unclear. Genetic predisposition, risk factors (2), relationships with the irritable bowel syndrome (3-5), a low-fibre diet, involvement of intestinal microbiota and the mucosal immune activation (6-7) remain elements whose significance is yet to be confirmed. The management, medical and surgical approach and the prevention of relapses of diverticular disease remain above all empirical and supported by few controlled clinical studies (8-9). This scenario of uncertainty may result in waste and diagnostic/therapeutic pathways not always suitable for a disease with such a high prevalence rate. On the basis of these considerations, there is a need to collect systematic information useful for determining aetiopathogenetic aspects and outcomes with greater accuracy.

OBJECTIVES OF THE STUDY

The purpose of the study is to structure a national register on an IT platform useful for determining:

1. The clinical aspects of diverticulosis/ diverticular disease
2. The risk factors of diverticulosis/ diverticular disease
3. The risk of complications of diverticular disease and the factors of risk and protection against complications.
4. The management of medical and surgical treatments

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients satisfying the following inclusion criteria are recruited:

1. Acceptance to sign the Informed Consent form
2. Age >18
3. Instrumental evidence (endoscopic or radiological) of diverticula in the colon.

Exclusion Criteria:

1. Refusal to sign the Informed Consent form
2. Inability to comply with the study procedures

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with colonic diverticula
Sampling Method: Non-Probability Sample
Enrollment: 1217 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Risk factors of diverticulosis/ diverticular disease | Five years
  Evaluation of demographic and clinical characteristics, including comorbidities and co-treatment, able to characterize the subgroups of patients with diverticular disease

SECONDARY OUTCOMES:
Risk of complications of diverticular disease and the factors of risk and protection against complications | Five years
  To evaluate risk factors for occurrence and recurrence of diverticulitis

OTHER OUTCOMES:
Clinical aspects of diverticulosis/ diverticular disease | Five years
  To evaluate clinical characteristics associated to diverticulosis, symptomatic uncomplicated diverticular disease and diverticulitis

REFERENCES:
- [Background] Annibale B, Lahner E, Maconi G, Usai P, Marchi S, Bassotti G, Barbara G, Cuomo R. Clinical features of symptomatic uncomplicated diverticular disease: a multicenter Italian survey. Int J Colorectal Dis. 2012 Sep;27(9):1151-9. doi: 10.1007/s00384-012-1488-5. Epub 2012 May 10. PMID 22573184
- [Background] Cuomo R, Barbara G, Andreozzi P, Bassotti G, Casetti T, Grassini M, Ierardi E, Maconi G, Marchi S, Sarnelli G, Savarino V, Usai P, Vozzella L, Annibale B. Symptom patterns can distinguish diverticular disease from irritable bowel syndrome. Eur J Clin Invest. 2013 Nov;43(11):1147-55. doi: 10.1111/eci.12152. Epub 2013 Sep 2. PMID 23992370
- [Background] Annibale B, Maconi G, Lahner E, De Giorgi F, Cuomo R. Efficacy of Lactobacillus paracasei sub. paracasei F19 on abdominal symptoms in patients with symptomatic uncomplicated diverticular disease: a pilot study. Minerva Gastroenterol Dietol. 2011 Mar;57(1):13-22. PMID 21372765
- [Background] Maconi G, Barbara G, Bosetti C, Cuomo R, Annibale B. Treatment of diverticular disease of the colon and prevention of acute diverticulitis: a systematic review. Dis Colon Rectum. 2011 Oct;54(10):1326-38. doi: 10.1097/DCR.0b013e318223cb2b. PMID 21904150
- [Background] Zullo A, Hassan C, Maconi G, Manes G, Tammaro G, De Francesco V, Annibale B, Ficano L, Buri L, Gatto G, Lorenzetti R, Campo SM, Ierardi E, Pace F, Morini S. Cyclic antibiotic therapy for diverticular disease: a critical reappraisal. J Gastrointestin Liver Dis. 2010 Sep;19(3):295-302. PMID 20922195
- [Derived] Carabotti M, Marasco G, Sbarigia C, Cuomo R, Barbara G, Pace F, Sarnelli G, Annibale B; at behalf of REMAD group. Site and duration of abdominal pain discriminate symptomatic uncomplicated diverticular disease from previous diverticulitis patients. Intern Emerg Med. 2024 Aug;19(5):1235-1245. doi: 10.1007/s11739-024-03588-6. Epub 2024 Apr 27. PMID 38671294
- [Derived] Cremon C, Carabotti M, Cuomo R, Pace F, Andreozzi P, Barbaro MR, Annibale B, Barbara G. Italian nationwide survey of pharmacologic treatments in diverticular disease: Results from the REMAD registry. United European Gastroenterol J. 2019 Jul;7(6):815-824. doi: 10.1177/2050640619845990. Epub 2019 Apr 20. PMID 31316786